CLINICAL TRIAL: NCT00469001
Title: Phase 1 Study of Using BNP as Guided Parameter in Treatment HF
Brief Title: Evaluation of NT PRO BNP Guided Therapy on Hospitalization Rate and Mortality in Patients With Chronic HF NYHA II-IY
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Other Study IDs: 00001
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Heart Failure
Keywords: Hospitalization and death from exacerbation CHF.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Treatment according NT Pro BNP level

SUMMARY:
To use continuous measurement of NT Pro BNP level as guide in therapy patients with CHF.

DETAILED DESCRIPTION:
Group of 100 patients with CHF, NYHA II-IY will be followed for 1 years in outpatient clinic of our hospital for hospitalization, death, 6 min walking protocol, number of decompensation as a primary end point. 50 patients will be treated according usual practice in outpatient clinics and in 50 patients will be additionally used level of NT Pro BNP as additional parameter.If level NT Pro BNP will be goes down will not be changes in treatment regiment. If level of NT Pro BNP will be increased treatment will be intensified.At the end of 1 year follow up we will compare the result of two strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patient older 18 y.old with CHF NYHA II-IY.

Exclusion Criteria:

* All conditions with life expectancy less than 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic heart failure. Half of the patients were treated by common medical practice for patients with heart failure. The other half were treated according to BNP values and common medical practice.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shochat, MD, PhD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel